CLINICAL TRIAL: NCT01590953
Title: A Study of the Effects of an Employee Wellness Program
Status: Completed | Type: Observational
Sponsor: Richard Deichmann, MD (Other)
Responsible Party: Sponsor-Investigator, Richard Deichmann, MD, PI, Ochsner Health System
Organization: Ochsner Health System (Other)
Other Study IDs: 2012.049.a
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ochsner employees with a body mass index (BMI) greater than or equal to 30 will be enrolled in a fitness program consisting 90 days of a structured exercise program and dietary counseling. Measures of fitness including weight, BMI, cholesterol, HDL, blood pressure, and absenteeism rates will be measured at 0, 90 days, in one year.

ELIGIBILITY:
Inclusion Criteria:

* Ochsner employees with a BMI greater than or equal to 30

Exclusion Criteria:

* Failure to pass initial physical exam

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ochsner employees with a BMI greater than or equal to 30
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2012-05-21 (Actual); Primary Completion 2014-05-21 (Actual); Study Completion 2014-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Elmwood fitness center, Harahan, Louisiana, United States